CLINICAL TRIAL: NCT06296927
Title: The Effect of the Emotional Freedom Technique Applied During Mammography Screening on Perceived Pain, Situational Anxiety and Satisfaction Levels
Brief Title: Effect of Emotional Freedom Technique on Perceived Pain, Situational Anxiety and Satisfaction Levels During Mammography Screening.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sümeyye Köse, Principal Investigator Midwife, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SumeyyeKose-E.138186
Record Dates: First submitted 2024-02-27; First posted 2024-03-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Mammography Screening; Pain; Anxiety
Keywords: mammography; pain; Emotional Freedom Technique
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled two-group study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Emotional Freedom Technique will be applied to women in the intervention group applying for mammography screening 30-40 minutes before the procedure.
  Interventions: Other: Emotional Freedom Technique
- Control Group (No Intervention): Women in the control group applying for mammography screening will not receive any intervention other than routine mammography screening.

INTERVENTIONS:
Other: Emotional Freedom Technique — The researcher will apply the Emotional Freedom Technique to women in the intervention group who apply for mammography screening for 30-40 minutes before the screening.
  Arms: Intervention Group

SUMMARY:
This study was planned to determine the effect of Emotional Freedom Technique on perceived pain level, situational anxietyl and satisfaction level during mammography screening.

DETAILED DESCRIPTION:
The randomized controlled and experimental study will be conducted with 94 women who applied to the Cancer Early Diagnosis, Screening and Education Center for mammography screening. The women in the experimental group (n=47) will be applied the Emotional Freedom Technique before mammography screening and the women in the control group (n=47) will be given routine mammography screening. The Sociodemographic Information Form, Visual Analog, Situational Anxiety Inventory, blood pressure monitor, thermometer and saturation device will be used to collect the data.

ELIGIBILITY:
Inclusion Criteria:

* Having a first mammography screening
* Knowing how to read and write,
* Having entered menopause (at least 1 year has passed since the last menstruation)

Exclusion Criteria:

* Having any cognitive or hearing problems,
* Having used painkillers before the procedure,
* Having no chronic diseases (cardiovascular, respiratory tract),
* Having a diagnosed mental illness (schizophrenia, bipolar disorder),
* Having epilepsy (as it is a contraindication for EFT applications),

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Anxiety | 20 minute
  Data will be collected using the State Anxiety Inventory. The answer options collected in four classes on the State Anxiety Inventory scale are: (1) Not at all, (2) A little, (3) A lot and (4) Completely; The options on the trait anxiety scale are (1) Rarel, (2) Sometimes, (3) A lot of the time, and (4) Almost always. The higher the score obtained from the scales, the higher the person's anxiety is. The total score obtained from the scale varies between 20-80, and 20-39 indicates a mild anxiety level, 40-59 indicates a medium anxiety level, 60-79 indicates a high anxiety level, and 80 points indicates a panic anxiety level.
Pain Level | 10 minute
  Data will be collected using the Visual Analogue Scale. Pain can be given a score between 0 and 10 on the scale.The higher the scale score, the greater the pain.

SECONDARY OUTCOMES:
Satisfaction Level | 10 minutes
  Data will be collected using the Visual Analog Scale. Satisfaction can be given a score between 0 and 10 on the scale. The higher the scale score, the higher the satisfaction level.
Blood Pressure | 5 minutes
  The data will be measured with a blood pressure monitor, and the average normal value in blood pressure measurement will be accepted as 120/80 mmHg.
Thermometer | 5 minutes
  Data will be measured from the forehead with a fever measuring device and the average normal value in body temperature measurement will be accepted as 36.5-37.5.
Saturation | 5 minutes
  Data will be measured from the fingertip with a saturation device and the average normal value of the measurement will be accepted as between 95-100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Pendik District Health Directorate Maternal Child Health and Family Planning Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No